CLINICAL TRIAL: NCT03786562
Title: The Effect of Intravenous Nalbuphine on Postoperative Nausea and Vomiting With Intrathecal Morphine in Abdominoplastic Surgery.
Brief Title: The Effect of Intravenous Nalbuphine on PONV With Intrathecal Morphine in Abdominoplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman A. Ismail, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01003060501
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-03

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Intrathecal Morphine
- Nalbuphine group (Active Comparator)
  Interventions: Drug: Intrathecal Morphine + Intravenous Nalbuphine

INTERVENTIONS:
Drug: Intrathecal Morphine — Group 1
  Arms: Placebo group
Drug: Intrathecal Morphine + Intravenous Nalbuphine — Group 2
  Arms: Nalbuphine group

SUMMARY:
How effectively intravenous nalbuphine can reduce the incidence of PONV after intrathecal administration of morphine in abdominoplastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominoplasty under spinal anesthesia
* American Society of Anesthesiologists (ASA) class I and II.

Exclusion Criteria:

* allergy to local anesthetics
* bleeding diatheses
* local infection or sepsis

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female undergoing abdominoplasty
Enrollment: 80 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 24 hours
  A verbal descriptive scale (VDS) was used to assess the severity of PONV. ( no nausea=0, severe nausea= 10)
  by postoperative nausea and vomiting scale which range (o no nasuea to 10 sever vomating).
  A verbal descriptive scale (VDS) was used to assess the severity of PONV .

SECONDARY OUTCOMES:
postoperative pain and puririts. | 24 hours
  Visual analogue scale (VAS) pain scores (no pain = 0, worst possible pain = 10).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt